CLINICAL TRIAL: NCT00000719
Title: A Trial of Alternating 2',3'-Dideoxycytidine and Zidovudine in the Treatment of Patients With Advanced HIV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 050; 11024 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To determine the long-term safety and tolerance of four alternating and two intermittent regimens of zidovudine ( AZT ) and 2',3'-dideoxycytidine ( zalcitabine; ddC ) in the treatment of patients with advanced HIV disease who have had to discontinue AZT because of true hematologic intolerance to standard reduced doses of AZT.

AIDS is a serious infectious disease caused by a new family of retrovirus which is spread primarily through sexual contact and administration of blood or blood products. Individuals who are infected with HIV could therefore benefit from therapy with an effective anti-AIDS virus agent. AZT and ddC have both been tested as antiviral agents and their potentially beneficial effects may be limited by time- and dose-dependent toxicity. A combination regimen using shorter courses of AZT and ddC might therefore be able to sustain treatment without producing toxicity. In addition, since the two drugs exhibit their major toxicity on different organ systems, cumulative or additive toxicity would not be expected.

DETAILED DESCRIPTION:
AIDS is a serious infectious disease caused by a new family of retrovirus which is spread primarily through sexual contact and administration of blood or blood products. Individuals who are infected with HIV could therefore benefit from therapy with an effective anti-AIDS virus agent. AZT and ddC have both been tested as antiviral agents and their potentially beneficial effects may be limited by time- and dose-dependent toxicity. A combination regimen using shorter courses of AZT and ddC might therefore be able to sustain treatment without producing toxicity. In addition, since the two drugs exhibit their major toxicity on different organ systems, cumulative or additive toxicity would not be expected.

There are six study regimens. Four of these are alternating regimens: A 2-week cycle consisting of 1 week of AZT followed by 1 week of ddC and an 8-week cycle consisting of 4 weeks of AZT followed by 4 weeks of ddC. All patients on alternating regimens will receive AZT alone at the standard dose orally every 4 hours for either 1 or 4 weeks. After the AZT is stopped, patients receive ddC orally every 4 hours for either 1 or 4 weeks, which completes a treatment cycle. One of two doses of ddC is studied in each alternating regimen. Both doses must be tested because the optimal dose cannot be inferred from tests that have already been done. AZT is administered first in the hope that AZT-mediated reduction of p24 antigen load may reduce the occurrence of acute ddC toxicity. Two intermittent regimens are also studied and are included to assess the contribution of each drug in the alternating regimens. One program consists of 1 week of AZT followed by 1 week of no drug. The other consists of 1 week of ddC followed by 1 week of no drug. Drug dosing continues for a total of 48 weeks unless toxicity develops. Patients who complete 48 weeks of therapy are followed for 4 additional weeks off therapy. Patients removed from study because of toxicity are followed for 4 weeks or until toxicity resolves. If study participants complete 48 weeks of therapy and meet criteria for efficacy, the study drug regimen may be continued for an additional 32 weeks. A 4 week wash-out period off drug will not be required for patients continuing on study. AMENDED 09/24/90 Drug dosing will be discontinued as of 11/30/90.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine at prophylactic doses, but its use is discouraged in persons without a history of Pneumocystis carinii pneumonia (PCP).
* Acyclovir for acute disseminated zoster.
* Maintenance doses of pyrimethamine, amphotericin, and pentamidine are allowed for patients who recover from toxoplasmosis, cryptococcosis, or pneumocystosis acquired after study entry.

Patients included in the study must have HIV infection confirmed by ELISA test and must have a documented history of at least 4 weeks of zidovudine (AZT) treatment.

* While hemoglobin at the start of AZT therapy must have been = or > 9.5 g/dl and granulocyte count = or > 1200 cells/mm3 at the start of AZT therapy, hematologic toxicity due to a reduced dose of AZT will be defined as:
* Hematologic toxicity must have occurred during a period when AZT was administered at = or < 600 mg/day for at least 2 weeks.
* There must have been no evidence of a cause for toxicity other than HIV infection and AZT use.
* Hematologic intolerance may have consisted of hemoglobin toxicity, granulocyte toxicity, or both.
* Recovery from hematologic toxicity must be manifested by the presence of a granulocyte count of > 1000 cells/mm3 and a hemoglobin of > 9.5 g/dl. without transfusions during the preceding 4 weeks. Patients must also have no significant bilateral symptoms of peripheral neuropathy, although all patients may have any degree of stable unilateral neurologic deficit. Up to 24 patients may have certain moderate bilateral abnormalities of peripheral neuropathy. AZT may not have been administered within 14 days prior to entering the study.

Prior Medication:

Required:

* A documented history of at least 4 weeks of zidovudine treatment which resulted in hematologic toxicity at reduced dose.
* Allowed but discouraged:
* A1-721.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Known active AIDS opportunistic infections.
* Known mycobacteremia, although cultures may be pending at the time of enrollment.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to entry into the study or with concurrent neoplasms other than KS, basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Significant malabsorption as manifested by steatorrhea with greater than 10 percent weight loss within the last 3 months.
* Diabetes.

Concurrent Medication:

Excluded:

* Experimental medications.
* Aspirin.
* Acetaminophen.
* Nonsteroidal anti-inflammatory agents should be minimized, with continuous use for > 72 hours discouraged.
* Chronic suppressive anti-infective therapy other than inhaled pentamidine and neurotoxic drugs should be avoided.
* Continuous therapy for > 7 days of acyclovir is prohibited except for the acute treatment of disseminated herpes zoster infection.

Patients with the following are excluded:

* Known mycobacteremia, although cultures may be pending at the time of enrollment.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to entry into the study or with concurrent neoplasms other than KS, basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Significant malabsorption as manifested by steatorrhea with greater than 10 percent weight loss within the last 3 months.
* Diabetes.
* Known active AIDS opportunistic infections. Patients must also have no significant bilateral symptoms of peripheral neuropathy, although all patients may have any degree of stable unilateral neurologic deficit. Up to 24 patients may have certain moderate bilateral abnormalities of peripheral neuropathy. AZT may not have been administered within 14 days prior to entering the study.

Prior Medication:

Excluded within 30 days of study entry:

* Any antiretroviral agents except zidovudine (AZT).
* Discouraged:
* A1-721.
* Pentamidine at prophylactic doses in persons without a history of Pneumocystis carinii pneumonia (PCP).

Active substance and/or alcohol abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Bozzette, Study Chair; D Richman, Study Chair
Locations (7):
- United States (7):
  - USC CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - University of Minnesota, ACTU, Minneapolis, Minnesota

REFERENCES:
- [Background] Lathey JL, Marschner IC, Kabat B, Spector SA. Deterioration of detectable human immunodeficiency virus serum p24 antigen in samples stored for batch testing. J Clin Microbiol. 1997 Mar;35(3):631-5. doi: 10.1128/jcm.35.3.631-635.1997. PMID 9041402
- [Background] Gries JM, Troconiz IF, Verotta D, Jacobson M, Sheiner LB. A pooled analysis of CD4 response to zidovudine and zalcitabine treatment in patients with AIDS and AIDS-related complex. Clin Pharmacol Ther. 1997 Jan;61(1):70-82. doi: 10.1016/S0009-9236(97)90183-1. PMID 9024175
- [Background] Fichtenbaum CJ, Clifford DB, Powderly WG. Risk factors for dideoxynucleoside-induced toxic neuropathy in patients with the human immunodeficiency virus infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Oct 1;10(2):169-74. doi: 10.1097/00042560-199510020-00009. PMID 7552481
- [Background] Bozzette SA, Richman DD. Salvage therapy for zidovudine-intolerant HIV-infected patients with alternating and intermittent regimens of zidovudine and dideoxycytidine. Am J Med. 1990 May 21;88(5B):24S-26S. doi: 10.1016/0002-9343(90)90418-d. PMID 2159706
- [Background] LeLacheur SF, Simon GL. Exacerbation of dideoxycytidine-induced neuropathy with dideoxyinosine. J Acquir Immune Defic Syndr (1988). 1991;4(5):538-9. PMID 1849990
- [Background] Bozzette S, Skowron G, Arrezo J, Spector SA, Pettinelli C, Richman DD. ACTG 050: alternating (alt) and intermittent (INT) ddc and AZT in the treatment of persons with advanced HIV infection and hematologic intolerance to AZT. Int Conf AIDS. 1990 Jun 20-23;6(3):192 (abstract no SB425)